CLINICAL TRIAL: NCT01879007
Title: Phase I Trial for Pharmacokinetic Characteristics of Factive 200mg Intravenous Formulation (Gemifloxacin 200mg) With Factive 320mg Tablet Formulation (Gemifloxacin 320mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-AACL006
Record Dates: First submitted 2013-06-04; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases | interventions — Gemifloxacin

ARMS (2):
- group 1 (Experimental): received one intravenous administration and one oral medication with interval of 1 week,
  Interventions: Drug: Factive® Tab / Factive IV
- group 2 (Experimental): received one oral administration and one intravenous medication with interval of 1 week
  Interventions: Drug: Factive® Tab / Factive IV

INTERVENTIONS:
Drug: Factive® Tab / Factive IV

SUMMARY:
This study seeks to compare the pharmacokinetic characteristics of Factive 200mg Intravenous Formulation (Gemifloxacin 200mg) with those of Factive 320mg Tablet Formulation (Gemifloxacin 320mg) and to explore possibility of clinical use of the IV formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Korean males between 19 and 45 years of age, weighing within 15% deviation of the ideal weight (CRC criteria) and residing in Korea (Appendix 4)
2. Applicants judged eligible as subject based on health exams (interview, blood pressure, 12-lead ECG, physical exam, blood and urine tests, and other screening tests) conducted not more than three weeks prior to administration (those with two or less clinically significant results)
3. Applicants who can take part in the whole process of clinical study
4. Applicants who sufficiently received explanation on the purpose and content of clinical study, characteristics of the investigational products, etc., before participating in the study and gave written consent to participate in the study voluntarily

Exclusion Criteria:

1. Applicants who exhibit symptoms suspected to be those of acute diseases prior to the start of the study
2. Clinically significant kidney disease or liver disease
3. Cardiovascular, respiratory, renal, endocrine system, hematology (hemorrhagic diathresis), digestive system (peptic ulcer), central nerve system, psychiatric disorder, or malignant tumors; chronic diseases that can influence the absorption, distribution, metabolism, or excretion of drugs
4. Applicants who have been on an abnormal diet, which can influence the absorption, distribution, metabolism, or excretion of drugs
5. Medical history of gastrointestinal resection except appendectomy
6. Applicants testing positive for hepatitis B antigen, hepatitis C antibody, or HIV antibody;
7. Clinically significant allergic diseases (excluding mild allergic rhinitis that does not require medication)
8. Known history of hypersensitivity to drugs
9. Known history of developing complications such as epilepsy or other convulsive diseases
10. Excessive consumption of caffeine and alcohol or heavy smoker
11. History of alcohol or drug abuse
12. Applicants who cannot take the standard meals provided by ASAN Medical Center(AMC)
13. Donation of whole or apheresis blood prior to the administration
14. Participation in other clinical study as subjects prior to the administration
15. Applicants who have taken prescription drugs prior to the administration or OTC(over-the-counter) drugs prior to the administration and for which such medications are judged by the principal investigator to have an influence on this study or on the safety of the subject
16. Applicants who are highly likely to take other medication during the study
17. Applicants who took medication that induces or inhibits drug-metabolizing enzymes such as barbiturates or consumed excessive amounts of alcohol less than 1 month prior to the administration
18. Medical history of meningitis, encephalitis, or brain injury
19. Difficulty in cooperating with researchers in proceeding with the study

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
AUC | Up to 48 hr
Cmax | Up to 48 hr
Tmax | Up to 48 hr
MRT | Up to 48 hr
CL | Up to 48 hr
Vss | Up to 48 hr
F | Up to 48 hr

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical center, Seoul, South Korea